CLINICAL TRIAL: NCT02657603
Title: Continuous Adductor Canal Block With a New Catheter - Primary Placement and Secondary Repositioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kai Henrik Wiborg Lange (Other)
Responsible Party: Sponsor-Investigator, Kai Henrik Wiborg Lange, Head Of Research, Hillerod Hospital, Denmark
Organization: Hillerod Hospital, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H-15016829
Record Dates: First submitted 2016-01-11; First posted 2016-01-18 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Pain
Keywords: Peripheral Nerve Blocks
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LAX insertion of catheter (Active Comparator): Lidocaine 10mg/ml, 15 ml injected into the adductor canal
  Interventions: Drug: Lidocaine; Procedure: LAX insertion of catheter
- SAX insertion of catheter (Active Comparator): Lidocaine 10mg/ml, 15 ml injected into the contralateral adductor canal
  Interventions: Drug: Lidocaine; Procedure: SAX insertion of catheter

INTERVENTIONS:
Drug: Lidocaine — Lidocaine injected through the new Catheter (LAX)
  Other Names: Lidocainehydrochlorid; Xylocaine
  Arms: LAX insertion of catheter
Drug: Lidocaine — Lidocaine injected through the new Catheter (SAX)
  Other Names: Lidocainehydrochlorid; Xylocaine
  Arms: SAX insertion of catheter
Procedure: LAX insertion of catheter — ultra sound guided cather insertion in the long axis (LAX) of the adductor canal
  Arms: LAX insertion of catheter
Procedure: SAX insertion of catheter — ultra sound guided cather insertion in the short axis (SAX) of the adductor canal
  Arms: SAX insertion of catheter

SUMMARY:
This is a single center, randomized, blinded trial in healthy volunteers. The volunteers will receive bilateral placement of the new catheter corresponding to the adductor canal. Each volunteer will have a catheter placed in the adductor canal in both legs. The catheters are randomized to be placed either in the long-axis or short-axis plane of the adductor canal. Both catheters will be injected with local analgesics (LA). Allocation will be blinded to the volunteer and the investigator assessing sensory function. The volunteers will be sent home with the catheter in situ and return the following day. Injection with LA is repeated and sensory function is tested again. Furthermore catheter position is determined with ultrasound during injection. If sensory function is not affected by injection of LA then the catheter is visualized with ultrasound and repositioned followed by a second injection of LA and subsequent assessment of sensory function

DETAILED DESCRIPTION:
3.2.1 Allocation concealment The volunteers are randomized using sealed opaque envelopes with a 1:1 ratio. The randomization defines which leg will be used for insertion of a catheter in the long-axis plane and which leg will be used for insertion in the short-axis plane of the adductor canal. The envelopes are prepared by health personnel with no relation to the study based on a computer-generated list.

3.2.2 Blinding Volunteers will be blinded to allocation. An opaque sterile draping will be used for insertion to prevent volunteers from observing the catheter insertion. After insertion the catheters will be covered with bandages to prevent unblinding of the volunteers. The investigator responsible for insertion of the catheters will leave the room after insertion and a separate assessor blinded to allocation will perform outcome assessments. On day 2 the investigator responsible for primary insertion will assess catheter position with ultra-sound (US), record a video for the assessors, injection of local anesthetics and cover the catheter in bandages. A separate blinded assessor will again perform the outcome assessment

3.2.3 Execution During catheter placement the volunteers are monitored using pulse oximetry and a secure intravenous access is obtained. A baseline sensory assessment is performed where cold sensation on the medial side of the lower leg is tested using alcohol swabs.

A peripheral nerve catheter will be inserted on each side under US guidance. This involves skin punctures at the site of insertion and at the exit site. To facilitate insertion the skin is locally infiltrated with lidocaine. Intravenous analgesia is provided if necessary (alfentanil 0.5mg/ml).

One catheter is inserted in the short-axis plane of the adductor canal using an in plane technique. The second catheter is inserted in the long-axis plane using a dynamic combination of in plane and out of plane techniques. 10ml of normal saline is used for hydro dissection in both catheters. When the catheters are in place 15 mL of LA (lidocaine 10mg/ml) is injected in each catheter. Distance from catheter orifice to artery is noted in the short axis group and distance from catheter orifice to fascia penetration is noted in the long axis group. After injection, the catheters are fixated to the skin with dressings.

Successful primary placement of the catheters will be tested 30 minutes after injection by a blinded investigator using a bilateral assessment of sensory function as described previously. Furthermore, cutaneous mapping is performed to assess affected cutaneous area.

Subsequently the volunteers are sent home with the catheter in situ and return the following day. The volunteers are instructed not to exercise -i.e. running, cycling, weight training etc.

On day 2 the catheter position is assessed with US during injection of LA and the distance from catheter orifice to artery/fascia is determined. A sensory assessment is performed. If there is no loss of cold sensation the catheter is registered as displaced and is therefore manually repositioned and injected with LA using US guidance. Assessment of cold sensation is repeated. Further, two investigators will independently watch a video clip of the injection procedure to assess whether the position is within the adductor canal. Total duration of participation for the individual volunteers will be 2 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age.
* ASA classification ≤ II. (ASA physical status classification system)
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Distance from skin to adductor canal above 4 cm
* Previous or ongoing surgery, pain or other disability of the investigated region resulting in sensory or neurologic deficits in the investigated region.
* Allergy to LA.
* Pregnancy (all female participants will be tested for urine hCG), breastfeeding, or unwilling to practice birth control during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Loss of cold sensation | 30 minutes after injection
  Loss of cold sensation after injection of Lidocaine(LA)

SECONDARY OUTCOMES:
Discomfort during day 1 | 1 day
  Rating on a scale from 1-10 overall, at rest and during activities and disturbance of sleep
Loss of cold sensation on day 2 - indicating correct position of the catheter on day 2 | 1 day after insertion
  loss of cold sensation on the medial part of the lower leg after LA injection on day 2
Interrater agreement between 2 assessors whether catheter is within the adductor canal assessed by US video. | 1 day
  cohen's kappa for interrater agreement between assessments
Displacement distance | 1 day
  Distance from catheter orifice to artery is noted in the short axis group and distance from catheter orifice to fascia penetration is noted in the long axis group
Loss of cold sensation after repositioning if found to be displaced - Indicating successful repositioning | 1 day
  loss of cold sensation on the medial part of the lower leg after LA injection after attempted repositioning

OTHER OUTCOMES:
Procedure time | 1 hour
  time used from penetration of skin to needle exit.
insertion attempts | 1 hour
  number of skin punctures for insertion
Affected skin area | 1 hour
  cutaneous mapping of the skin area on the medial part of the lower with loss of cold sensation evaluated by application of an ice roller and outlining with a marker (pen) for comparison

CONTACTS AND LOCATIONS:
Overall Officials: Tobias S Lyngeraa, MD, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Nordsjællands Hospital, Hillerød, Denmark